CLINICAL TRIAL: NCT00657150
Title: A Phase III Randomised, Parallel Group, Double-blind, Active Controlled Study to Investigate the Efficacy and Safety of Orally Administered 220 mg Dabigatran Etexilate Capsules (110 mg Administered on the Day of Surgery Followed by 220 mg Once Daily) Compared to Subcutaneous 40 mg Enoxaparin Once Daily for 28-35 Days, in Prevention of Venous Thromboembolism in Patients With Primary Elective Total Hip Arthroplasty Surgery. (RE-NOVATE II)
Brief Title: Dabigatran Etexilate Compared With Enoxaparin in Prevention of Venous Thromboembolism (VTE) Following Total Hip Arthroplasty
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 1160.64; 2007-002630-11 (EudraCT Number: EudraCT)
Record Dates: First submitted 2008-03-27; First posted 2008-04-14 (Estimated); Results first posted 2010-12-17 (Estimated); Last update posted 2014-07-02 (Estimated); Status verified 2013-12

CONDITIONS: Venous Thromboembolism
MeSH Terms: conditions — Venous Thromboembolism | interventions — Enoxaparin; Dabigatran

ARMS (2):
- Dabigatran etexilate (Experimental): 220 mg once daily
  Interventions: Drug: Dabigatran etexilate
- Enoxaparin (Active Comparator): 40 mg once daily
  Interventions: Drug: Enoxaparin

INTERVENTIONS:
Drug: Enoxaparin — 40 mg once daily
  Arms: Enoxaparin
Drug: Dabigatran etexilate — 220 mg once daily
  Arms: Dabigatran etexilate

SUMMARY:
The primary objective of the trial is to demonstrate non-inferiority of 220 mg oral dabigatran etexilate compared to 40 mg subcutaneous enoxaparin administered once daily. Safety and efficacy will be compared between the treatment groups.

ELIGIBILITY:
Inclusion criteria:

* Patients scheduled to undergo primary, unilateral, elective total hip arthroplasty.
* Male or female 18 years of age or older.
* Patients giving written informed consent for study participation.

Exclusion criteria:

* Patients weighing less than 40 kg.
* History of bleeding diathesis.
* Patients who in the investigators judgement are perceived as having an excessive risk of bleeding, for example, constitutional or acquired coagulation disorders or because of anticipated need of quinidine, verapamil or other restricted medication during the treatment period (see Section 4.2.2).
* Major surgery or trauma (e.g., hip fracture) within 3 months of enrolment.
* Recent unstable cardiovascular disease (in the investigators opinion) such as uncontrolled hypertension, that is ongoing at the time of enrolment or history of myocardial infarction within 3 months of enrolment.
* Any history of haemorrhagic stroke or any of the following intracranial pathologies: bleeding, neoplasm, Atriovenous (AV) malformation or aneurysm.
* Ongoing treatment for Venous Thromboembolism (VTE).
* Clinically relevant bleeding (gastrointestinal, pulmonary, intraocular or urogenital bleeding) within 6 months of enrolment.
* Gastric or duodenal ulcer within one year of enrolment.
* Liver disease expected to have any potential impact on survival (ie, hepatitis B or C, cirrhosis). This does not include Gilberts syndrome or hepatitis A with complete recovery.
* Active liver disease or liver disease decreasing survival (e.g, acute hepatitis, chronic active hepatitis, cirrhosis) or Alanine Aminotransferase (ALT) >3 x ULN.
* Known severe renal insufficiency (CrCl <30 ml/min). Note: CrCl should be calculated only if serum creatinine is elevated or renal insufficiency is suspected. See Appendix 10.1 for calculation.
* Elevated creatinine that, in the investigators opinion, contraindicates venography.
* Treatment with anticoagulants, clopidogrel, ticlopidine, abciximab, aspirin >162.5 mg/day or NSAID with t 1/2 >12 hours within 7 days prior to hip replacement surgery OR anticipated need while the patient is receiving study medication and prior to 24 hours after the last administration of any blinded study medication (COX-2 selective inhibitors are allowed).
* Anticipated required use of intermittent pneumatic compression and electric stimulation of lower limb.
* Pre-menopausal women (last menstruation within 1 year prior to signing informed consent) who:

  * Are pregnant.
  * Are nursing.
  * Are of child-bearing potential and are NOT practicing acceptable methods of birth control, or do NOT plan to continue practicing an acceptable method throughout the study. Acceptable methods of birth control include intrauterine device; oral, implantable or injectable contraceptives and surgical sterility.
* Known allergy to radio opaque contrast media.
* History of thrombocytopenia, including heparin-induced thrombocytopenia, or a platelet count <100,000 cells/microliter at randomisation.
* Allergy to heparins or dabigatran etexilate.
* Active malignant disease or current cytostatic treatment. Patients should be disease free for at least 5 years.
* Participation in a clinical trial within 30 days of randomisation.
* Leg amputee.
* Known alcohol or drug abuse which would interfere with completion of the study.
* Contraindications to enoxaparin.
* Previous participation in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2055 (Actual)
Dates: Start 2008-03; Primary Completion 2009-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (108):
- United States (10):
  - 1160.64.01005 Boehringer Ingelheim Investigational Site, La Jolla, California
  - 1160.64.01010 Boehringer Ingelheim Investigational Site, Aurora, Colorado
  - 1160.64.01009 Boehringer Ingelheim Investigational Site, Englewood, Colorado
  - 1160.64.01012 Boehringer Ingelheim Investigational Site, Clearwater, Florida
  - 1160.64.01006 Boehringer Ingelheim Investigational Site, Lexington, Kentucky
  - 1160.64.01003 Boehringer Ingelheim Investigational Site, Missoula, Montana
  - 1160.64.01007 Boehringer Ingelheim Investigational Site, Charleston, South Carolina
  - 1160.64.01013 Boehringer Ingelheim Investigational Site, Conway, South Carolina
  - 1160.64.01002 Boehringer Ingelheim Investigational Site, Houston, Texas
  - 1160.64.01011 Boehringer Ingelheim Investigational Site, Spokane, Washington
- Australia (4):
  - 1160.64.2003 Boehringer Ingelheim Investigational Site, Daws Park, South Australia
  - 1160.64.2002 Boehringer Ingelheim Investigational Site, Box Hill, Victoria
  - 1160.64.2001 Boehringer Ingelheim Investigational Site, Windsor, Victoria
  - 1160.64.2004 Boehringer Ingelheim Investigational Site, Nedlands, Western Australia
- Austria (4):
  - 1160.64.4004 Boehringer Ingelheim Investigational Site, Graz
  - 1160.64.4002 Boehringer Ingelheim Investigational Site, Linz
  - 1160.64.4001 Boehringer Ingelheim Investigational Site, Vienna
  - 1160.64.4003 Boehringer Ingelheim Investigational Site, Wels
- Belgium (4):
  - 1160.64.5004 Boehringer Ingelheim Investigational Site, Brussels
  - 1160.64.5002 Boehringer Ingelheim Investigational Site, Deurne
  - 1160.64.5005 Boehringer Ingelheim Investigational Site, Lanaken
  - 1160.64.5001 Boehringer Ingelheim Investigational Site, Leuven
- Canada (10):
  - 1160.64.6009 Boehringer Ingelheim Investigational Site, Edmonton, Alberta
  - 1160.64.6002 Boehringer Ingelheim Investigational Site, Red Deer, Alberta
  - 1160.64.6012 Boehringer Ingelheim Investigational Site, Ajax, Ontario
  - 1160.64.6003 Boehringer Ingelheim Investigational Site, Belleville, Ontario
  - 1160.64.6004 Boehringer Ingelheim Investigational Site, Cambridge, Ontario
  - 1160.64.6008 Boehringer Ingelheim Investigational Site, Kitchener, Ontario
  - 1160.64.6011 Boehringer Ingelheim Investigational Site, Oshawa, Ontario
  - 1160.64.6005 Boehringer Ingelheim Investigational Site, Sarnia, Ontario
  - 1160.64.6007 Boehringer Ingelheim Investigational Site, Stratford, Ontario
  - 1160.64.6013 Boehringer Ingelheim Investigational Site, Windsor, Ontario
- Czechia (5):
  - 1160.64.7004 Boehringer Ingelheim Investigational Site, Chomutov
  - 1160.64.7005 Boehringer Ingelheim Investigational Site, Jihlava
  - 1160.64.7003 Boehringer Ingelheim Investigational Site, Kolín
  - 1160.64.7001 Boehringer Ingelheim Investigational Site, Pilsen
  - 1160.64.7002 Boehringer Ingelheim Investigational Site, Prague
- Denmark (4):
  - 1160.64.8004 Boehringer Ingelheim Investigational Site, Frederiksberg
  - 1160.64.8003 Boehringer Ingelheim Investigational Site, Herlev
  - 1160.64.8001 Boehringer Ingelheim Investigational Site, Hørsholm
  - 1160.64.8002 Boehringer Ingelheim Investigational Site, Silkeborg
- Finland (3):
  - 1160.64.9002 Boehringer Ingelheim Investigational Site, Jyväskylä
  - 1160.64.9001 Boehringer Ingelheim Investigational Site, Oulu
  - 1160.64.9003 Boehringer Ingelheim Investigational Site, Tampere
- Germany (4):
  - 1160.64.1104 Boehringer Ingelheim Investigational Site, Garmisch-Partenkirchen
  - 1160.64.1101 Boehringer Ingelheim Investigational Site, Mainz
  - 1160.64.1103 Boehringer Ingelheim Investigational Site, Markgröningen
  - 1160.64.1102 Boehringer Ingelheim Investigational Site, Rheinfelden
- Hungary (4):
  - 1160.64.1201 Boehringer Ingelheim Investigational Site, Gyula
  - 1160.64.1203 Boehringer Ingelheim Investigational Site, Kecskemét
  - 1160.64.1202 Boehringer Ingelheim Investigational Site, Szeged
  - 1160.64.1204 Boehringer Ingelheim Investigational Site, Székesfehérvár
- India (13):
  - 1160.64.9105 Boehringer Ingelheim Investigational Site, Ahmedabad
  - 1160.64.9112 Boehringer Ingelheim Investigational Site, Andhra Pradesh
  - 1160.64.9109 Boehringer Ingelheim Investigational Site, Andhra Predesh
  - 1160.64.9103 Boehringer Ingelheim Investigational Site, Bangalore
  - 1160.64.9108 Boehringer Ingelheim Investigational Site, Bangalore
  - 1160.64.9107 Boehringer Ingelheim Investigational Site, Baroda
  - 1160.64.9110 Boehringer Ingelheim Investigational Site, Mangalore
  - 1160.64.9104 Boehringer Ingelheim Investigational Site, Mohali
  - 1160.64.9111 Boehringer Ingelheim Investigational Site, New Delhi
  - 1160.64.9106 Boehringer Ingelheim Investigational Site, Pune
  - 1160.64.9101 Boehringer Ingelheim Investigational Site, Ramdaspeth Nagpur
  - 1160.64.9102 Boehringer Ingelheim Investigational Site, Secunderabad
  - 1160.64.9113 Boehringer Ingelheim Investigational Site, Vadodara
- Italy (6):
  - 1160.64.1401 Boehringer Ingelheim Investigational Site, Bologna
  - 1160.64.1405 Boehringer Ingelheim Investigational Site, Parma
  - 1160.64.1402 Boehringer Ingelheim Investigational Site, Pavia
  - 1160.64.1407 Boehringer Ingelheim Investigational Site, Reggio Emilia
  - 1160.64.1403 Boehringer Ingelheim Investigational Site, Roma
  - 1160.64.1404 Boehringer Ingelheim Investigational Site, Torino
- Netherlands (7):
  - 1160.64.1503 Boehringer Ingelheim Investigational Site, Amsterdam
  - 1160.64.1507 Boehringer Ingelheim Investigational Site, Amsterdam
  - 1160.64.1501 Boehringer Ingelheim Investigational Site, Hilversum
  - 1160.64.1506 Boehringer Ingelheim Investigational Site, Hoofddorp
  - 1160.64.1510 Boehringer Ingelheim Investigational Site, Leiden
  - 1160.64.1505 Boehringer Ingelheim Investigational Site, Sittard
  - 1160.64.1508 Boehringer Ingelheim Investigational Site, Zwolle
- 1160.64.3001 Boehringer Ingelheim Investigational Site, Takapuna Auckland, New Zealand
- Norway (5):
  - 1160.64.1603 Boehringer Ingelheim Investigational Site, Ålesund
  - 1160.64.1601 Boehringer Ingelheim Investigational Site, Bodø
  - 1160.64.1606 Boehringer Ingelheim Investigational Site, Elverum
  - 1160.64.1604 Boehringer Ingelheim Investigational Site, Lillehammer
  - 1160.64.1605 Boehringer Ingelheim Investigational Site, Tynset
- Poland (5):
  - 1160.64.1702 Boehringer Ingelheim Investigational Site, Krakow
  - 1160.64.1704 Boehringer Ingelheim Investigational Site, Krakow
  - 1160.64.1705 Boehringer Ingelheim Investigational Site, Lodz
  - 1160.64.1703 Boehringer Ingelheim Investigational Site, Piekary Śląskie
  - 1160.64.1701 Boehringer Ingelheim Investigational Site, Warsaw
- South Africa (3):
  - 1160.64.1801 Boehringer Ingelheim Investigational Site, Bryanston
  - 1160.64.1804 Boehringer Ingelheim Investigational Site, Cape Western Province
  - 1160.64.1802 Boehringer Ingelheim Investigational Site, Plumstead
- Spain (6):
  - 1160.64.1904 Boehringer Ingelheim Investigational Site, Alcorcón (Madrid)
  - 1160.64.1906 Boehringer Ingelheim Investigational Site, Barcelona
  - 1160.64.1908 Boehringer Ingelheim Investigational Site, Fuenlabrada
  - 1160.64.1901 Boehringer Ingelheim Investigational Site, Madrid
  - 1160.64.1907 Boehringer Ingelheim Investigational Site, Madrid
  - 1160.64.1905 Boehringer Ingelheim Investigational Site, Valencia
- Sweden (10):
  - 1160.64.2101 Boehringer Ingelheim Investigational Site, Gothenburg
  - 1160.64.2112 Boehringer Ingelheim Investigational Site, Halmstad
  - 1160.64.2105 Boehringer Ingelheim Investigational Site, Hässleholm
  - 1160.64.2109 Boehringer Ingelheim Investigational Site, Kalmar
  - 1160.64.2103 Boehringer Ingelheim Investigational Site, Kungälv
  - 1160.64.2106 Boehringer Ingelheim Investigational Site, Lidköping
  - 1160.64.2102 Boehringer Ingelheim Investigational Site, Motala
  - 1160.64.2108 Boehringer Ingelheim Investigational Site, Stockholm
  - 1160.64.2111 Boehringer Ingelheim Investigational Site, Uppsala
  - 1160.64.2107 Boehringer Ingelheim Investigational Site, Varberg

REFERENCES:
- [Derived] Eriksson BI, Dahl OE, Rosencher N, Clemens A, Hantel S, Feuring M, Kreuzer J, Huo M, Friedman RJ. Oral dabigatran etexilate versus enoxaparin for venous thromboembolism prevention after total hip arthroplasty: pooled analysis of two phase 3 randomized trials. Thromb J. 2015 Nov 17;13:36. doi: 10.1186/s12959-015-0067-8. eCollection 2015. PMID 26578849
- [Derived] Eriksson BI, Dahl OE, Huo MH, Kurth AA, Hantel S, Hermansson K, Schnee JM, Friedman RJ; RE-NOVATE II Study Group. Oral dabigatran versus enoxaparin for thromboprophylaxis after primary total hip arthroplasty (RE-NOVATE II*). A randomised, double-blind, non-inferiority trial. Thromb Haemost. 2011 Apr;105(4):721-9. doi: 10.1160/TH10-10-0679. Epub 2011 Jan 12. PMID 21225098

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The treatment period is from first administration of study medication, until 3 days after last administration of study medication. Treatment duration is planned for 28 - 35 days. The study period is from first administration of study medication until day 84 - 91.
Pre-assignment Details: Whilst 2055 patients were randomised to treatment prior to surgery in this trial, only 2013 started treatment. Therefore, 42 patients were randomised but not treated.
Groups:
- Dabigatran 220mg: qd (once daily) oral
- Enoxaparin: 40mg qd (once daily) subcutaneous
Period: Overall Study
Arm/Group | Dabigatran 220mg | Enoxaparin
Started | 1010 | 1003
Completed | 895 | 910
Not Completed | 115 | 93
Not completed — Adverse Event | 19 | 10
Not completed — Non-compliant with protocol | 5 | 9
Not completed — Lost to Follow-up | 2 | 0
Not completed — Withdrawal by Subject | 51 | 36
Not completed — Other | 38 | 38
Period: Treatment
Arm/Group | Dabigatran 220mg | Enoxaparin
Started | 1010 | 1003
Completed | 903 | 906
Not Completed | 107 | 97
Not completed — Adverse Event | 60 | 53
Not completed — Non-compliant with protocol | 10 | 9
Not completed — Lost to Follow-up | 1 | 0
Not completed — Withdrawal by Subject | 23 | 20
Not completed — Other | 13 | 15

BASELINE CHARACTERISTICS:
Population: Treated set
Groups:
- Total: Total of all reporting groups
Arm/Group | Dabigatran 220mg | Enoxaparin | Total
Number analyzed (Participants) | 1010 | 1003 | 2013
Age, Continuous [Mean (Standard Deviation); unit: Years] | 61.9 (11.5) | 62.0 (11.3) | 62.0 (11.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 541 | 501 | 1042
  Male | 469 | 502 | 971
Body Mass Index N=(1003;992;1995) [Mean (Standard Deviation); unit: kg/m^2] | 27.8 (4.8) | 27.8 (4.8) | 27.8 (4.8)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Total Venous Thromboembolic Event and All-cause Mortality During Treatment Period
Description: Total Venous Thromboembolic Event (VTE) includes both proximal and distal deep vein thrombosis (DVT) (detected by routine venography), symptomatic DVT (confirmed by venous duplex, ultrasound, venography or autopsy) and pulmonary embolism (PE) (confirmed by pulmonary V-Q scintigraphy, chest x-ray, pulmonary angiography, spiral CT or autopsy).
  All of these components and all deaths were centrally adjudicated by the VTE events committee, which was not aware of the treatment allocation of the patients.
Time Frame: 28-35 days
Population: Full Analysis Set (randomised, had taken at least 1 dose of oral or subcutaneous trial medication, had undergone surgery, had evaluable negative venogram for both distal and proximal DVT in both legs or positive venography in any 1 segment of 1 or both legs, or confirmed symptomatic DVT, PE or death during the treatment period.)
Measure: Number; unit: Participants
Arm/Group | Dabigatran 220mg | Enoxaparin
Number analyzed (Participants) | 792 | 786
Participants | 61 | 69
Statistical Analysis 1: Comparison: Dabigatran 220mg vs Enoxaparin; Risk difference versus Enoxaparin; Test type: Non-Inferiority or Equivalence — Non-inferiority Analysis with NI margin 7.7%; p < 0.0001, Normal approximation — Superiority p-value = 0.4367; Normal approximation of independent binomial distribution without stratification; Risk Difference (Percentage) = -1.08, 95% CI [-3.79 to 1.64]

2. Secondary Outcome: Number of Participants With Major Venous Thromboembolic Event and Venous Thromboembolic Event-related Mortality During Treatment Period
Description: Major Venous Thromboembolic Event (VTE) is defined as proximal DVT and PE, as adjudicated by the VTE events committee
Time Frame: 28-35 days
Population: Full Analysis Set-major (randomised, had taken at least 1 dose of oral or subcutaneous trial medication, had undergone surgery, had evaluable negative venogram for proximal DVT in both legs or a positive venogram for proximal DVT in either leg or confirmed symptomatic proximal DVT, PE or death related to VTE during the treatment period.)
Measure: Number; unit: Participants
Arm/Group | Dabigatran 220mg | Enoxaparin
Number analyzed (Participants) | 805 | 795
Participants | 18 | 33
Statistical Analysis 1: Comparison: Dabigatran 220mg vs Enoxaparin; Test type: Superiority or Other; p = 0.029, Normal approximation; Normal approximation of independent binomial distribution without stratification; Risk Difference (RD) = -1.91, 95% CI [-3.64 to -0.19]

3. Secondary Outcome: Number of Participants With Proximal Deep Vein Thrombosis During Treatment Period
Description: Proximal Deep Vein Thrombosis as adjudicated by the VTE events committee
Time Frame: 28-35 days
Population: Full Analysis Set - pDVT (all patients who had been randomised, had taken at least 1 dose of oral or subcutaneous trial medication, had undergone surgery (i.e. a date of surgery was reported), evaluable negative venogram for proximal DVT in both legs or positive venogram in either leg or confirmed symptomatic proximal DVT)
Measure: Number; unit: Participants
Arm/Group | Dabigatran 220mg | Enoxaparin
Number analyzed (Participants) | 804 | 793
Participants | 17 | 31
Statistical Analysis 1: Comparison: Dabigatran 220mg vs Enoxaparin; Risk difference versus Enoxaparin; Test type: Superiority or Other; p = 0.0358, Normal approximation; Normal approximation of independent binomial distribution without stratification; Risk Difference (Percentage) = -1.79, 95% CI [-3.47 to -0.12]

4. Secondary Outcome: Number of Participants With Total Deep Vein Thrombosis During Treatment Period
Description: Total Deep Vein Thrombosis as adjudicated by the VTE events committee
Time Frame: 28-35 days
Population: Full Analysis Set-tDVT (randomised, had taken at least 1 dose of oral or subcutaneous trial medication, had undergone surgery, evaluable negative venogram for both distal and proximal DVT in both legs or positive venography in any 1 segment of 1 or both legs, or confirmed symptomatic DVT.)
Measure: Number; unit: Participants
Arm/Group | Dabigatran 220mg | Enoxaparin
Number analyzed (Participants) | 791 | 784
Participants | 60 | 67
Statistical Analysis 1: Comparison: Dabigatran 220mg vs Enoxaparin; Risk difference versus Enoxaparin; Test type: Superiority or Other; p = 0.4839, Normal approximation; Normal approximation of independent binomial distribution without stratification; Risk Difference (Percentage) = -0.96, 95% CI 2-sided [-3.65 to 1.73]

5. Secondary Outcome: Number of Participants With Symptomatic Deep Vein Thrombosis During Treatment Period
Description: Symptomatic Deep Vein Thrombosis, confirmed by venous duplex, ultrasound, venography or autopsy, and as adjudicated by the VTE events committee
Time Frame: 28-35 days
Population: Full Analysis Set - op (all patients who had been randomised, had taken at least 1 dose of oral or subcutaneous trial medication or had undergone surgery (i.e. a date of surgery was reported)
Measure: Number; unit: Participants
Arm/Group | Dabigatran 220mg | Enoxaparin
Number analyzed (Participants) | 1001 | 992
Participants | 0 | 4
Statistical Analysis 1: Comparison: Dabigatran 220mg vs Enoxaparin; Comparison versus Enoxaparin; Test type: Superiority or Other; p = 0.0612, Fisher Exact

6. Secondary Outcome: Number of Participants With Pulmonary Embolism During Treatment Period
Description: Pulmonary embolism confirmed by pulmonary V-Q scintigraphy, chest x-ray, pulmonary angiography, spiral CT or autopsy, and as adjudicated by the VTE events committee
Time Frame: 28-35 days
Population: as for outcome 5
Measure: Number; unit: Participants
Arm/Group | Dabigatran 220mg | Enoxaparin
Number analyzed (Participants) | 1001 | 992
Participants | 1 | 2
Statistical Analysis 1: Comparison: Dabigatran 220mg vs Enoxaparin; Comparison versus Enoxaparin; Test type: Superiority or Other; p = 0.6231, Fisher Exact

7. Secondary Outcome: Number of Participants Who Died During Treatment Period
Description: All cause death, as adjudicated by the VTE events committee
Time Frame: 28-35 days
Population: as for outcome 5
Measure: Number; unit: Participants
Arm/Group | Dabigatran 220mg | Enoxaparin
Number analyzed (Participants) | 1001 | 992
Participants | 0 | 1
Statistical Analysis 1: Comparison: Dabigatran 220mg vs Enoxaparin; Comparison versus Enoxaparin; Test type: Superiority or Other; p = 0.4977, Fisher Exact

8. Secondary Outcome: Number of Participants With Total Venous Thromboembolic Event (VTE) and All-cause Mortality During the Follow-up Period
Description: Total Venous Thromboembolic Event (VTE) includes both proximal and distal deep vein thrombosis (DVT) (detected by routine venography), symptomatic DVT (confirmed by venous duplex, ultrasound, venography or autopsy) and pulmonary embolism (PE) (confirmed by pulmonary V-Q scintigraphy, chest x-ray, pulmonary angiography, spiral CT or autopsy).
Time Frame: 3 months
Population: Patients with any data available during follow-up
Measure: Number; unit: Participants
Arm/Group | Dabigatran 220mg | Enoxaparin
Number analyzed (Participants) | 942 | 951
Participants
  Total VTE and all-cause mortality | 2 | 4
  asymptomatic Deep Vein Thrombosis | 0 | 1
  symptomatic Deep Vein Thrombosis | 1 | 0
  Pulmonary Embolism | 1 | 2
  death | 0 | 1
Statistical Analysis 1: Comparison: Dabigatran 220mg vs Enoxaparin; Comparison versus Enoxaparin; Test type: Superiority or Other; p = 0.6870, Fisher Exact

9. Secondary Outcome: Number of Participants With Bleeding Events (Defined According to Modified McMaster Criteria) During Treatment Period
Description: Major bleeding events were defined as
  * fatal
  * clinically overt associated with loss of haemoglobin >=20g/L in excess of what was expected
  * clinically overt leading to the transfusion of >=2 units packed cells or whole blood in excess of what was expected
  * symptomatic retroperitoneal, intracranial, intraocular or intraspinal
  * requiring treatment cessation
  * leading to re-operation
  Clinically-relevant was defined as
  * spontaneous skin hematoma >=25 cm²
  * wound hematoma >=100 cm²
  * spontaneous nose bleed >5 min
  * macroscopic hematuria spontaneous or >24 hours if associated with an intervention
  * spontaneous rectal bleeding
  * gingival bleeding >5 min
  * any other bleeding event considered clinically relevant by the investigator
  Any bleeding events were defined as major, clinically-relevant and minor bleeding events. Minor bleeding events were defined as all other bleeding events that did not fulfil the criteria from above.
Time Frame: 28-35 days
Population: All patients who had been randomised, had taken at least 1 dose of oral or subcutaneous trial medication.
Measure: Number; unit: Participants
Arm/Group | Dabigatran 220mg | Enoxaparin
Number analyzed (Participants) | 1010 | 1003
Participants
  Major bleeding events | 14 | 9
  Major and clinically relevant bleeding events | 37 | 29
  Any bleeding events | 98 | 83
Statistical Analysis 1: Comparison: Dabigatran 220mg vs Enoxaparin; Comparison versus Enoxaparin for the category major bleeding events; Test type: Superiority or Other; p = 0.4022, Fisher Exact
Statistical Analysis 2: Comparison: Dabigatran 220mg vs Enoxaparin; Absolute difference versus Enoxaparin for the category major and clinically relevant bleeding events; Test type: Superiority or Other; p = 0.3305, Normal approximation; Normal approximation of independent binomial distribution; Absolute Difference (Percentage) = 0.8, 95% CI 2-sided [-0.8 to 2.3]
Statistical Analysis 3: Comparison: Dabigatran 220mg vs Enoxaparin; Absolute difference versus Enoxaparin for the category any bleeding events; Test type: Superiority or Other; p = 0.2626, Normal approximation; Normal approximation of independent binomial distribution; Absolute Difference (Percentage) = 1.4, 95% CI 2-sided [-1.1 to 3.9]

10. Secondary Outcome: Blood Transfusion
Description: Number of treated and operated patients with required blood transfusion on day of surgery.
Time Frame: Day 1
Population: Treated and operated patients
Measure: Number; unit: participants
Arm/Group | Dabigatran 220mg | Enoxaparin
Number analyzed (Participants) | 1001 | 992
participants
  Transfusions required | 246 | 237
  Missing | 4 | 7

11. Secondary Outcome: Volume of Blood Loss
Description: Volume of blood loss for treated and operated patients during surgery.
Time Frame: Day 1
Population: Treated and operated patients
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | Dabigatran 220mg | Enoxaparin
Number analyzed (Participants) | 967 | 957
mL | 404.9 (259.67) | 411.0 (275.38)

12. Secondary Outcome: Laboratory Analyses
Description: Frequency of patients with possible clinically significant abnormalities.
Time Frame: First administration to end of study
Population: Treated patients
Measure: Number; unit: participants
Arm/Group | Dabigatran 220mg | Enoxaparin
Number analyzed (Participants) | 966 | 962
participants
  AST increase N=(964;962) | 28 | 44
  AST decrease N=(964;962) | 0 | 0
  ALT increase N=(966;962) | 34 | 67
  ALT decrease N=(966;962) | 0 | 0
  Bilirubin increase N=(966;962) | 3 | 1
  Bilirubin decrease N=(966;962) | 0 | 0

ADVERSE EVENTS:
Time Frame: 31 - 38 days
Description: Treatment emergent events (last medication + 3 days)
Arm/Group | Dabigatran 220mg | Enoxaparin
Serious Adverse Events (participants affected / at risk) | 57/1010 | 59/1003
Other Adverse Events (participants affected / at risk) | 389/1010 | 389/1003
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Dabigatran 220mg (N=1010) | Enoxaparin (N=1003)
Anaemia (Blood and lymphatic system disorders) | 1 | 0
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 1 | 0
Thrombocytosis (Blood and lymphatic system disorders) | 1 | 0
Atrial fibrillation (Cardiac disorders) | 1 | 1
Cardiac arrest (Cardiac disorders) | 2 | 0
Cardiac failure congestive (Cardiac disorders) | 0 | 1
Myocardial infarction (Cardiac disorders) | 1 | 1
Supraventricular tachycardia (Cardiac disorders) | 1 | 0
Retinal artery occlusion (Eye disorders) | 0 | 1
Abdominal distension (Gastrointestinal disorders) | 0 | 1
Abdominal hernia (Gastrointestinal disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 1
Anal haemorrhage (Gastrointestinal disorders) | 0 | 1
Constipation (Gastrointestinal disorders) | 0 | 2
Gastric ulcer (Gastrointestinal disorders) | 0 | 1
Ileus (Gastrointestinal disorders) | 0 | 1
Ileus paralytic (Gastrointestinal disorders) | 0 | 1
Intestinal obstruction (Gastrointestinal disorders) | 1 | 1
Intestinal perforation (Gastrointestinal disorders) | 1 | 0
Melaena (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 2
Oesophageal perforation (Gastrointestinal disorders) | 0 | 1
Oesophagitis (Gastrointestinal disorders) | 0 | 1
Rectal haemorrhage (Gastrointestinal disorders) | 2 | 0
Vomiting (Gastrointestinal disorders) | 0 | 2
Asthenia (General disorders) | 1 | 0
Hyperthermia (General disorders) | 0 | 1
Impaired healing (General disorders) | 0 | 1
Inflammation (General disorders) | 1 | 1
Multi-organ failure (General disorders) | 1 | 0
Oedema peripheral (General disorders) | 1 | 1
Pyrexia (General disorders) | 2 | 0
Secretion discharge (General disorders) | 1 | 0
Cholelithiasis (Hepatobiliary disorders) | 1 | 0
Abscess neck (Infections and infestations) | 0 | 1
Arthritis infective (Infections and infestations) | 0 | 2
Diverticulitis (Infections and infestations) | 0 | 1
Haematoma infection (Infections and infestations) | 1 | 0
Hepatitis A (Infections and infestations) | 1 | 0
Injection site abscess (Infections and infestations) | 0 | 1
Oesophageal candidiasis (Infections and infestations) | 1 | 0
Post procedural infection (Infections and infestations) | 1 | 0
Postoperative wound infection (Infections and infestations) | 1 | 1
Urinary tract infection (Infections and infestations) | 0 | 2
Wound infection (Infections and infestations) | 2 | 0
Abdominal injury (Injury, poisoning and procedural complications) | 1 | 0
Avulsion fracture (Injury, poisoning and procedural complications) | 1 | 0
Brain contusion (Injury, poisoning and procedural complications) | 1 | 0
Device dislocation (Injury, poisoning and procedural complications) | 1 | 0
Dislocation of joint prosthesis (Injury, poisoning and procedural complications) | 2 | 0
Fat embolism (Injury, poisoning and procedural complications) | 1 | 0
Femur fracture (Injury, poisoning and procedural complications) | 2 | 3
Fracture (Injury, poisoning and procedural complications) | 0 | 1
Genital injury (Injury, poisoning and procedural complications) | 1 | 0
Hip fracture (Injury, poisoning and procedural complications) | 0 | 1
Joint dislocation (Injury, poisoning and procedural complications) | 4 | 3
Oesophageal injury (Injury, poisoning and procedural complications) | 0 | 1
Operative haemorrhage (Injury, poisoning and procedural complications) | 2 | 0
Periprosthetic fracture (Injury, poisoning and procedural complications) | 0 | 2
Post procedural discharge (Injury, poisoning and procedural complications) | 1 | 0
Post procedural haematoma (Injury, poisoning and procedural complications) | 0 | 1
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 2 | 0
Procedural hypotension (Injury, poisoning and procedural complications) | 0 | 1
Seroma (Injury, poisoning and procedural complications) | 0 | 1
Traumatic haematoma (Injury, poisoning and procedural complications) | 1 | 1
Wound dehiscence (Injury, poisoning and procedural complications) | 0 | 1
Wound haemorrhage (Injury, poisoning and procedural complications) | 1 | 1
Wound secretion (Injury, poisoning and procedural complications) | 3 | 1
C-reactive protein increased (Investigations) | 1 | 0
Haemoglobin decreased (Investigations) | 1 | 0
Hepatic enzyme increased (Investigations) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 1
Metabolic acidosis (Metabolism and nutrition disorders) | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Haemarthrosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Joint effusion (Musculoskeletal and connective tissue disorders) | 0 | 1
Mobility decreased (Musculoskeletal and connective tissue disorders) | 0 | 1
Carotid artery stenosis (Nervous system disorders) | 0 | 1
Central nervous system lesion (Nervous system disorders) | 0 | 1
Epilepsy (Nervous system disorders) | 1 | 0
Monoparesis (Nervous system disorders) | 0 | 1
Somnolence (Nervous system disorders) | 1 | 0
Syncope (Nervous system disorders) | 1 | 1
Transient ischaemic attack (Nervous system disorders) | 2 | 0
Anuria (Renal and urinary disorders) | 1 | 0
Renal failure acute (Renal and urinary disorders) | 0 | 4
Renal impairment (Renal and urinary disorders) | 0 | 1
Urethral stenosis (Renal and urinary disorders) | 0 | 1
Urinary retention (Renal and urinary disorders) | 1 | 0
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 1
Hip arthroplasty (Surgical and medical procedures) | 1 | 0
Deep vein thrombosis (Vascular disorders) | 4 | 10
Haemorrhage (Vascular disorders) | 1 | 0
Shock haemorrhagic (Vascular disorders) | 1 | 0
Thrombophlebitis superficial (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Dabigatran 220mg (N=1010) | Enoxaparin (N=1003)
Constipation (Gastrointestinal disorders) | 100 | 102
Nausea (Gastrointestinal disorders) | 162 | 166
Vomiting (Gastrointestinal disorders) | 110 | 94
Pyrexia (General disorders) | 62 | 80
Haemoglobin decreased (Investigations) | 56 | 62
Hypotension (Vascular disorders) | 61 | 51

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Any publication of the result of this trial must be consistent with the Boehringer Ingelheim publication policy. The rights of the investigator and of the sponsor with regard to publication of the results of this trial are described in the investigator contract.